CLINICAL TRIAL: NCT00715988
Title: Safety and Single Dose Population Pharmacokinetics and Bioavailability of Methadone and Its Enantiomers in Newborns and Young Infants At 29-48 Weeks Post Menstrual Age
Brief Title: Methadone Pharmacokinetics and Cardiac Effects in Newborns
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Case Western Reserve University (Other); Children's Mercy Hospital Kansas City (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Robert Ward, Professor, Pediatrics; Adjunct Professor, Pharmacology/Toxicology, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24569; 1U10HD045986-01 (NIH)
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Pain
Keywords: Methadone; analgesia; newborns; QT prolongation; Young Infants
MeSH Terms: conditions — Pain; Agnosia; Long QT Syndrome | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Scheme 1 (Experimental): Patients who are feeding or not feeding and mechanically ventilated, >/=3 d of age and 29 0/7wks-48 6/7 wks PMA, treated with i.v. bolus doses or infusion of fentanyl, morphine or methadone for clinical indications, with arterial/venous line in place & expected treatment for at least 1-2 more days. Pk sampling = 0.5 ml blood samples x6/infant. ECG monitoring. Three patients will be enrolled in 5 PMA groups. Should apnea or hypotension occur, dosages for Treatment Scheme 2 will be reduced (50%); more patients will be studied in Treatment Scheme 1 to insure that the lower dose is well tolerated & effective.
  Interventions: Drug: Methadone
- Scheme 2 (Experimental): Patients defined in Scheme 1, tolerating feeds for >/= 3 days will be studied twice, after i.v. methadone and after enteral methadone after the end of sampling after the first dose. 4-5 samples will be obtained after dose 1 and after dose 2 depending on PMA and weight. Patients will be divided into groups based on PMA..
  Interventions: Drug: Methadone HCl Inject 10 mg/ml (will require dilution)

INTERVENTIONS:
Drug: Methadone HCl Inject 10 mg/ml (will require dilution) — Methadone HCl oral solution 5 mg/ml Methadone HCl inject 10 mg/ml (will require dilution)
  Other Names: Dolophine, Methadose, Methadose Oral
  Arms: Scheme 2
Drug: Methadone — Methadone HCl oral solution 5 mg/ml Methadone HCl inject 10 ml/ml (will require dilution) Single dose
  Other Names: Dolophine, Methadose, Methadose Oral
  Arms: Scheme 1

SUMMARY:
The Primary objectives of this proposal are to determine the population kinetics for methadone and its enantiomers in preterm newborns and infants at 29 weeks to 48 weeks post menstrual age (PMA) who are 1 week old and older and establish any correlations of the kinetics with PMA to determine the bioavailability for enterally administered methadone in these newborns and young infants.

The secondary objectives of this proposal are to explore possible genotypic changes in CYP3A4-3A7-3A5, CYP2B6, CYP2C8, CYP2C19, and CYP2D6 and PGO on the kinetics of methadone in neonates and young infants and to test the safety of methadone in this population by correlating the plasma concentrations of the methadone enantiomers, S-methadone and R-methadone, with changes in cardiac repolarization by measurement of corrected QT, heart rate, and blood pressure.

DETAILED DESCRIPTION:
Painful procedures are frequent during the NICU care of sick newborns. Newborns are capable of perceiving pain by the time in fetal development when they reach our current limits of viability around 23-24 weeks post menstrual age.1 Painful procedures include suctioning during mechanical ventilation, thoracostomy tube placement, heel lance and venipuncture for blood sampling, and care following surgical procedures such as PDA ligation and bowel resection. Simons et al recently reported on the number of painful procedures in a large NICU in Rotterdam and provided a review of the frequency of such procedures from other NICU's.2 This review shows that before discharge from the NICU, newborns may experience as many as 376 painful procedures and as many as 61 painful procedures in a single day (or more if all procedures were not observed or reported). The most frequent procedures were heel lance and suctioning, both associated with the need for mechanical ventilation. Topical treatment of pain from heel lance has not been successful with EMLA3 or tetracaine.4

During initial NICU care for infants supported with mechanical ventilation, systemic analgesia is usually provided with parenteral treatment with fentanyl or morphine. Most neonates are extubated soon after birth, and continued systemic treatment with analgesics is not needed. Other neonates have problems associated with chronic pain or continued painful procedures, such as surgical problems, chronic lung disease, airway anomalies, pulmonary hypoplasia and pulmonary hypertension following ECMO and congenital diaphragmatic hernia repair. These patients often require mechanical ventilation for weeks and sometimes months. During that prolonged care, systemic analgesia is changed to enteral dosing to reduce risks of infection associated with central catheters and to reduce the number of intravenous catheter insertions.

Morphine and fentanyl administered enterally do not provide reliable systemic concentrations and effects due to first-pass metabolism. Fentanyl undergoes first-pass metabolism by CYP3A4 during passage through the intestines and liver. Morphine undergoes first pass hepatic metabolism primarily by UGT2B7. In addition for morphine, one of its major metabolites, the 3-glucuronide, is anti-analgesic and can cause dysphoria. An effective and well-characterized systemic analgesic that can be administered enterally is needed for the care of infants who require prolonged analgesic treatment and methadone can meet those needs.

Methadone treatment in adults provides effective systemic analgesia after enteral administration through binding to the mu opioid receptor with a wide range of reported half-lives of 5 to 130 hrs,5 2 to 50 hrs,6 and 33 to 46 hrs; 7 and bioavailability ranging from 41 to 95%.8, 9

Recently, methadone was reported to prolong QTc in adults receiving large doses of methadone during chronic treatment, often with additional predisposing factors for QT prolongation. Methadone is dispensed in a racemic mixture whose enantiomers have different potency for analgesia and for binding to the myocardium to potentially prolong QT. In addition the different enantiomers exhibit complex kinetics in adults as they undergo metabolism, primarily by CYP3A4, CYP2B6, and CYP2C19. This study will evaluate kinetics and bioavailability of methadone enantiomers and its effects on QT of neonates and young infants.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients must be in the NICU or PICU with continuous cardiorespiratory monitoring
2. PMA between 29 0/7 to 48 6/7 weeks (EGA at birth (wks) + postnatal age wks) at the start of study
3. Weight >1499 gm at the time of enrollment
4. Postnatal age of 3 days or more
5. Arterial or venous catheter suitable for blood sampling with a separate i.v. infusion site is preferred, but not essential
6. Currently being treated with methadone bolus doses or fentanyl or morphine in bolus doses or by infusion for clinical indications and expected to be treated for at least 1-2 more days with opioids for study of single dose pharmacokinetics and to be treated for 3-5 days more during the study of bioavailability
7. Hematocrit ≥35%
8. Parental permission
9. Approval by the patient's attending physician

   Treatment Scheme 1, studied for 48 hr after a single i.v. dose of methadone
10. Feeding or not feeding
11. Mechanically ventilated

    Treatment Scheme 2 studied for 24 to 48 hr after a single i.v. dose of methadone AND again after a single enteral dose of methadone after the end of sampling after the first dose; order of doses is randomized. If the caregiver feels the patient is too sedated at the end of pK sampling after Dose, 1, then Dose 2 will be delayed until patient is judged to need analgesic treatment.
12. Tolerating enteral feeding for 3 consecutive days before study

EXCLUSION CRITERIA

1. Clinically diagnosed liver dysfunction
2. Clinically diagnosed kidney dysfunction with urine output <1.0 ml/kg/hr
3. Gastrointestinal malformation or dysfunction that might interfere with enteral drug absorption
4. Congenital anomalies or other conditions thought to be incompatible with life
5. History of arrhythmias, excluding bradycardia associated with apnea
6. Unstable cardiorespiratory status
7. Serum K+ <3.0 mEq/L
8. QTc[H] >0.449 ms using Hodges correction =QT + 1.75(rate - 60).
9. Family history of unexplained early cardiac deaths, syncope, or long QT syndrome in primary relatives: siblings, parents, grandparents, or aunts/uncles.
10. Treatment with inhibitors and inducers of CYP3A4, CYP2B6, CYP2D6 and PGP including:

amiodarone, carbamazepine, ciprofloxacin, clarithromycin, clotrimazole, dexamethasone, erythromycin, ethosuximide, fluconazole, fluoxetine, fluvoxamine, grapefruit juice, indinavir, itraconazole, ketoconazole, metronidazole, miconazole, nelfinavir, paroxetine, phenobarbital, phenytoin, quercetin, quinidine, rifabutin, rifampin, ritonavir, saquinavir, sulfadimidine, sulfinpyrazone, troleandomycin

Ages: 29 Weeks to 48 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2007-10; Primary Completion 2012-09 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
Find the population kinetics for methadone and its enantiomers in preterm newborns and infants at 29 weeks to 48 wks PMA who are 1 week old and older | 48 hours

SECONDARY OUTCOMES:
Measure the effects of R and S enantiomers of methadone on QT interval in newborns | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ward, M.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data shared with other investigators leading to publication of the pediatric population pharmacokinetics of methadone

REFERENCES:
- [Derived] Ward RM, Drover DR, Hammer GB, Stemland CJ, Kern S, Tristani-Firouzi M, Lugo RA, Satterfield K, Anderson BJ. The pharmacokinetics of methadone and its metabolites in neonates, infants, and children. Paediatr Anaesth. 2014 Jun;24(6):591-601. doi: 10.1111/pan.12385. Epub 2014 Mar 26. PMID 24666686